CLINICAL TRIAL: NCT02381379
Title: A Randomized Control Trial Comparing Peginterferon-α-2a Versus Observation After Stopping Tyrosine Kinase Inhibitor in Chronic Myeloid Leukemia With Deep Molecular Response for at Least Two Years
Brief Title: Malaysia Stop Tyrosine Kinase Inhibitor Trial
Acronym: MSIT
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ministry of Health, Malaysia (Other Government)
Responsible Party: Principal Investigator, Dr Kuan Jew Win, Dr, Ministry of Health, Malaysia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NMRR-13-1186-15491
Record Dates: First submitted 2015-03-02; First posted 2015-03-06 (Estimated); Last update posted 2020-09-14 (Actual); Status verified 2020-09

CONDITIONS: Leukemia, Chronic Myeloid
Keywords: CML; peginterferon; stop; BCR-ABL
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — peginterferon alfa-2a

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Peginterferon-α-2a (Pegasys®) (Active Comparator): Subcutaneous peginterferon-α-2a (PEGASYS®) starting at 180µg weekly for one year
  Interventions: Drug: Peginterferon-α-2a
- Observation (No Intervention): Stop tyrosine kinase inhibitor that was on and no active medication that might affect CML, for example any immune-modulatory agents, traditional herbs or medications, chemotherapeutic agents, growth factors, or colony stimulating factors is allowed during the trial period.

INTERVENTIONS:
Drug: Peginterferon-α-2a — Subcutaneous peginterferon-α-2a (PEGASYS®) starting at 180µg weekly for one year.
  Other Names: Pegasys®
  Arms: Peginterferon-α-2a (Pegasys®)

SUMMARY:
To compare administration of peginterferon-α-2a for 1 year versus observation after stopping tyrosine kinase inhibitor (TKI) in chronic myeloid leukemia (CML) patients with deep MR ≥ 2 years.

DETAILED DESCRIPTION:
Chronic myeloid leukemia (CML) is a chronic myeloproliferative neoplasm signified by the presence of Philadephia chromosome, which is the derivative of chromosome 22 after translocation between chromosome 9 and 22. The Philadephia chromosome will produce the mutated tyrosine kinase (BCR-ABL1), which will initiate the pathogenesis of the disease.

Imatinib is the first tyrosine kinase inhibitor (TKI), which has changed the treatment paradigm of CML since its approval from U.S. Food and Drug Administration in 2001 for the treatment of CML. It signifies a new era of oncological treatment using targeted therapy. Subsequent generation TKIs have been marketed as a more potent therapy for CML. Tyrosine kinase inhibitor is conventionally thought not able to cure CML and it has to be taken for life. It is able to induce a very deep molecular response (MR) in about 10% of CML patients as evidenced by persistent undetectable or ≤0.0032% (International Scale IS) BCR-ABL1 transcript in quantitative polymerase chain reaction (PCR) test on current molecular assays, which is labelled as MR4.5 or more. However these patients have to continue taking their TKIs as per recommendations from the European Leukaemia Net and this is the current practice in our institution and in Malaysia. Long term treatment is cumbersome, there is a concern of chronic side effects with long term tyrosine kinase inhibition and it is a financial burden on most countries' health budget as these drugs are very expensive.

Current available data showed that 40% of CML patients with prior stable MR4.5 for 2 years or more will be able to stay imatinib-free for at least 2 years. About 13% of patients without confirmed molecular relapse by the study criteria have low persistent BCR-ABL1 but remain imatinib-free for median follow-up of 22 months (range 6 - 35). A few patients with confirmed molecular relapse by study criteria remained drug free on follow-up. This postulates a component of immunity suppressing the leukemic clone.

Interferon is the standard treatment of CML before the era of TKI. As a single agent, it induces complete cytogenetic response (CCR) in about 20%, and non-sustainable deep MR in about 10% of patients in early chronic phase. These are much smaller figures compared to TKI. Imatinib at the dose of 400mg daily induces CCR in about 70% and deep MR in about 10% of patient in chronic phase after one year of treatment. However, interferon-responded patients may indeed retain the response once interferon was withdrawn via interferon-induced immunity towards the leukemic clone, which leads to longer drug free period compared to TKI. Hence, it is logical to postulate the use of interferon after TKI was stopped when patients have attained deep MR for more than two years will increase the percentage of patients remain TKI-free on follow-up. Unfortunately, there are not many studies concerning this matter. Carella et al described a case series of five patients with deep MR ranging from 12 to 41 months, were put on interferon with follow-up ranging from three to 16 months. Recently, there was a study from Japan, nine out of 12 analyzable patients including 3 patients with previous treatment of interferon, who stopped TKI, was put on interferon remained in deep MR after median follow-up of 23 months (6-27 months). In regards to peginterferon, there is a small studies by Hardan I et al describing 11 CML patients with various responses after imatinib (from complete cytogenetic response N=3, major molecular response N=6, deep MR N=2) were put on peginterferon-α-2a for nine months together with imatinib, then imatinib was stopped and continued with peginterferon-α-2a for another three months. It is difficult to draw any conclusion from this paper because of the small number of subjects, only two subjects have achieved deep MR (with unknown duration) before study entry, and peginterferon-α-2a was combined with imatinib for nine months which will cloud the true effect of peginterferon-α-2a after imatinib was stopped.

So far, there is no randomized study comparing interferon administered for fix duration after TKI was stopped versus observation to see whether the percentage and duration of CML patient who remains TKI-free can be increased and prolonged with interferon, respectively. It will be of interest to see how long the group which was given interferon remains TKI-free. If they remain TKI-free for a long duration, it not only suggests the interferon-induced immunity, but also suggests the interferon-induced immunity can be induced when only a very low level of leukemic cells present. Economical wise, TKI-free certainly give a big relief on the limited health budget of the on-growing CML population.

ELIGIBILITY:
Inclusion Criteria:

* The subject must be 18 years old or above
* The subject has CML in chronic phase during diagnosis
* The subject is treated with ongoing TKI at any dose for at least 3 years
* The subject has achieved stable deep molecular response (DMR) on International Scale (IS) for 2 years or more by any TKI
* Definition of deep molecular response (IS) ≥ 2 years

  * Deep molecular response = MR4 (IS 0.01%) or better
  * There must be at least 2 results (including the latest) of MR4.5 with an acceptable control gene copy number for the assay over the last two years
  * There must not be any result exceeding a major molecular response (MMR) (IS 0.1%) over the last two years
* The latest PCR result should be compelled with Intervention Start Date, which is within 4 weeks of Study Entry Date or 17 weeks of the latest PCR test.

Exclusion Criteria:

* The subject has previous history of any TKI failure as according to European LeukemiaNet 2009(17).
* The subject has previous history of successfully engrafted autologous or allogeneic haematopoeitic stem cell transplant and after transplant no disease relapse as defined by MSIT protocol
* The subject is planned for autologous or allogeneic stem cell transplantation
* The subject has previous history of interferon or peginterferon administration and achieved complete cytogenetic response with interferon or peginterferon
* The subject had undergone or on immune-modulatory treatments other than interferon or peginterferon
* The subject is undergoing treatment for other malignancies
* The subject has haemoglobin <9g/dL and platelet count <90x109/L for two successive readings of 1 month apart
* The subject has positive Hepatitis B surface Ag (HBsAg), Hepatitis C antibody (anti-HCV), or Human Immunodeficiency Virus 1 antibody (anti-HIV1)
* The subject has creatinine clearance of ≤50mL/min
* The subject has persistent alanine transaminase ≥2x upper normal limit for two successive readings of 1 month apart.
* Adults under law protection or without ability to consent
* The subject has previous history or on-going psychiatric illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Estimated)
Dates: Start 2015-03 (Actual); Primary Completion 2018-10 (Actual); Study Completion 2021-10 (Estimated)

PRIMARY OUTCOMES:
Relapse rate | 3 years
  Relapse is defined as either i. Loss of MMR, which is a reading of > 0.1% IS, which need to be confirmed by a second analysis point if no previous increasing trend of PCR result, or ii. Positivity of BCR-ABL1 transcripts in quantitative PCR, as confirmed by a second analysis point, indicating the increase (at least 1 log) in relation to the first analysis point at two successive assessments.

SECONDARY OUTCOMES:
The number of patients who developed adverse side-effects of interferon | 1 year
  The number of patients who developed adverse side-effects of interferon vs observation arm.
The rate of reattaining deep MR | 3 years
  The success rate of reattaining deep MR after restarting TKI in those patients who relapse.
Time to regain deep MR after relapse | 3 years
  Defined as time of relapse to the first time point, after restarting whatever treatment, patient has deep MR confirmed by second analysis point.
Quality of life (QoL) assessment | 3 year
  Assessed by questionnaire from INTERNATIONAL PROJECT ON QUALITY OF LIFE IN CHRONIC MYELOID LEUKEMIA.

CONTACTS AND LOCATIONS:
Overall Officials: Kian Meng Chang, FRCP(London), Principal Investigator — Ampang Hospital, Malaysia
Locations (9):
- Malaysia (9):
  - Sultanah Aminah Hospital, Johor Bahru, Johor
  - Sultanah Bahiyah Hospital, Alor Star, Kedah
  - Queen Elizabeth Hospital, Kota Kinabalu, Sabah
  - Sarawak General Hospital, Kuching, Sarawak
  - Miri Hospital, Miri, Sarawak
  - Sibu Hospital, Sibu, Sarawak
  - Ampang Hospital, Ampang, Selangor
  - Malacca General Hospital, Malacca
  - Hospital Pulau Pinang, Pulau Pinang

REFERENCES:
- [Background] Mahon FX, Rea D, Guilhot J, Guilhot F, Huguet F, Nicolini F, Legros L, Charbonnier A, Guerci A, Varet B, Etienne G, Reiffers J, Rousselot P; Intergroupe Francais des Leucemies Myeloides Chroniques. Discontinuation of imatinib in patients with chronic myeloid leukaemia who have maintained complete molecular remission for at least 2 years: the prospective, multicentre Stop Imatinib (STIM) trial. Lancet Oncol. 2010 Nov;11(11):1029-35. doi: 10.1016/S1470-2045(10)70233-3. Epub 2010 Oct 19. PMID 20965785
- [Background] Ross DM, Branford S, Seymour JF, Schwarer AP, Arthur C, Bartley PA, Slader C, Field C, Dang P, Filshie RJ, Mills AK, Grigg AP, Melo JV, Hughes TP. Patients with chronic myeloid leukemia who maintain a complete molecular response after stopping imatinib treatment have evidence of persistent leukemia by DNA PCR. Leukemia. 2010 Oct;24(10):1719-24. doi: 10.1038/leu.2010.185. Epub 2010 Sep 2. PMID 20811403
- [Background] Kantarjian HM, O'Brien S, Cortes JE, Shan J, Giles FJ, Rios MB, Faderl SH, Wierda WG, Ferrajoli A, Verstovsek S, Keating MJ, Freireich EJ, Talpaz M. Complete cytogenetic and molecular responses to interferon-alpha-based therapy for chronic myelogenous leukemia are associated with excellent long-term prognosis. Cancer. 2003 Feb 15;97(4):1033-41. doi: 10.1002/cncr.11223. PMID 12569603
- [Background] Preudhomme C, Guilhot J, Nicolini FE, Guerci-Bresler A, Rigal-Huguet F, Maloisel F, Coiteux V, Gardembas M, Berthou C, Vekhoff A, Rea D, Jourdan E, Allard C, Delmer A, Rousselot P, Legros L, Berger M, Corm S, Etienne G, Roche-Lestienne C, Eclache V, Mahon FX, Guilhot F; SPIRIT Investigators; France Intergroupe des Leucemies Myeloides Chroniques (Fi-LMC). Imatinib plus peginterferon alfa-2a in chronic myeloid leukemia. N Engl J Med. 2010 Dec 23;363(26):2511-21. doi: 10.1056/NEJMoa1004095. PMID 21175313
- [Background] Verbeek W, Konig H, Boehm J, Kohl D, Lange C, Heuer T, Scheibenbogen C, Reis HE, Hochhaus A, Graeven U. Continuous complete hematological and cytogenetic remission with molecular minimal residual disease 9 years after discontinuation of interferon-alpha in a patient with Philadelphia chromosome-positive chronic myeloid leukemia. Acta Haematol. 2006;115(1-2):109-12. doi: 10.1159/000089476. PMID 16424660
- [Background] Mahon FX, Delbrel X, Cony-Makhoul P, Faberes C, Boiron JM, Barthe C, Bilhou-Nabera C, Pigneux A, Marit G, Reiffers J. Follow-up of complete cytogenetic remission in patients with chronic myeloid leukemia after cessation of interferon alfa. J Clin Oncol. 2002 Jan 1;20(1):214-20. doi: 10.1200/JCO.2002.20.1.214. PMID 11773172
- [Background] Usuki K, Kanda Y, Iijima K, Iki S, Hirai H, Urabe A. [Chronic myelogenous leukemia in cessation of therapy after sustained CCR with interferon]. Rinsho Ketsueki. 2003 Dec;44(12):1161-5. Japanese. PMID 14978932
- [Background] Mauro E. Long-term molecular response after discontinuation of interferon-alpha in two patients with chronic myeloid leukaemia. Blood Transfus. 2012 Oct;10(4):559; author reply 560. doi: 10.2450/2012.0144-11. Epub 2012 Feb 29. No abstract available. PMID 22395358
- [Background] Veneri D, Tecchio C, De Matteis G, Paviati E, Benati M, Franchini M, Pizzolo G. Long-term persistence of molecular response after discontinuation of interferon-alpha in two patients with chronic myeloid leukaemia. Blood Transfus. 2012 Apr;10(2):233-4. doi: 10.2450/2011.0057-11. Epub 2011 Sep 22. No abstract available. PMID 22044951
- [Background] Hardan I, Stanevsky A, Volchek Y, Tohami T, Amariglio N, Trakhtenbrot L, Koren-Michowitz M, Shimoni A, Nagler A. Treatment with interferon alpha prior to discontinuation of imatinib in patients with chronic myeloid leukemia. Cytokine. 2012 Feb;57(2):290-3. doi: 10.1016/j.cyto.2011.11.018. Epub 2011 Dec 13. PMID 22169779
- [Background] Carella AM. Interferon-alpha is able to maintain complete molecular remission induced by imatinib after its discontinuation. Leukemia. 2008 May;22(5):1090-1. doi: 10.1038/leu.2008.94. Epub 2008 Apr 3. No abstract available. PMID 18385749
- [Background] Baccarani M, Cortes J, Pane F, Niederwieser D, Saglio G, Apperley J, Cervantes F, Deininger M, Gratwohl A, Guilhot F, Hochhaus A, Horowitz M, Hughes T, Kantarjian H, Larson R, Radich J, Simonsson B, Silver RT, Goldman J, Hehlmann R; European LeukemiaNet. Chronic myeloid leukemia: an update of concepts and management recommendations of European LeukemiaNet. J Clin Oncol. 2009 Dec 10;27(35):6041-51. doi: 10.1200/JCO.2009.25.0779. Epub 2009 Nov 2. PMID 19884523